CLINICAL TRIAL: NCT00801242
Title: An Open-Label, Multi-Centre, Uncontrolled, Trial Investigating Degarelix One-Month Dosing Regimen Administered as Intermittent Androgen Deprivation (IAD) for One or More Cycles in Patients With Prostate Cancer Requiring Androgen Deprivation Therapy
Brief Title: Intermittent Treatment With Degarelix of Patients Suffering From Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS29; 2008-003931-19 (EudraCT Number)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix 240 mg / 80 mg (Experimental)
  Interventions: Drug: Degarelix 240 mg / 80 mg

INTERVENTIONS:
Drug: Degarelix 240 mg / 80 mg — For each treatment cycle, a starting dose of 240 mg of degarelix was administered on Day 0 as two 120 mg subcutaneous (s.c.) injections in the abdominal region. Thereafter, 6 doses of 80 mg degarelix were administered 28 days apart via single s.c. injections.
  Other Names: FE200486; Firmagon

SUMMARY:
The purpose of this uncontrolled, multi-center, open-label trial was to investigate the feasibility of using degarelix as intermittent androgen deprivation (IAD) therapy in the treatment of prostate cancer.

DETAILED DESCRIPTION:
The participants received one or more treatment cycles of seven monthly degarelix doses during the induction period(s). The off-treatment period(s) started when prostate-specific antigen (PSA) ≤4 ng/mL and lasted up to 24 months based on PSA levels. A visit was scheduled on a monthly basis during the induction treatment periods, and every two months during the off-treatment periods. During the off-treatment periods, degarelix treatment was re-initiated when PSA >4 ng/mL. The maximum of degarelix IAD treatment cycles that a participant could receive was limited to three.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent before any trial-related activity is performed. A trial-related activity is defined as any procedure that would not have been performed during the normal management of the patient.
* Has a histologically confirmed (Gleason graded) adenocarcinoma of the prostate (all stages), and is in need of androgen deprivation treatment.
* Patients with Locally Advanced or Metastatic Prostate Cancer - Screening PSA level (measured at a central laboratory) must be >4 ng/mL and ≤50 ng/mL.
* Patients with Localised Prostate Cancer or Patients with Previous Therapy with Curative Intention and a Rising PSA - PSA doubling time (based on patient records at the trial site) must be <24 months. There is no minimum PSA level required and the maximum PSA must be ≤50 ng/mL.
* Is a male patient aged 18 years or older.
* Has an Eastern Cooperative Oncology Group score of ≤2.
* Has a life expectancy of at least 24 months.

Exclusion Criteria:

* Has had previous or is currently under hormonal management of prostate cancer (surgical castration or other hormonal manipulation, including gonadotropin releasing hormone (GnRH) receptor agonists, GnRH antagonists, anti-androgens, 5-alpha reductase inhibitors and estrogens). However, for patients having undergone prostatectomy or radiotherapy with curative intention, then neoadjuvant/adjuvant hormonal therapy for a maximum duration of 6 months is accepted. This treatment should have been terminated at least 6 months prior to Screening Visit.
* Is considered to be candidate for curative therapy, i.e. radical prostatectomy or radiotherapy.
* Has a history of severe uncontrolled asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Has hypersensitivity towards any component of the investigational medicinal product.
* Has had cancer within the last five years except prostate cancer and surgically removed basal or squamous cell carcinoma of the skin.
* Has a known or suspected clinically significant liver and/or biliary disease.
* Has a history of or risk factors for Torsades de Pointes
* At time of inclusion receives concomitant medications that might prolong the QT interval.
* Has any clinically significant laboratory abnormalities which in the judgment of the investigator would affect the patient's health or the outcome of the trial.
* Has a clinically significant disorder (other than prostate cancer) including but not limited to renal, haematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease, and alcohol or drug abuse or any other condition, which may affect the patient's health or the outcome of the trial as judged by the investigator.
* Has severe kidney failure (creatinine clearance <30 mL/min), based on the serum creatinine value at Screening Visit and calculated by Cockcroft-Gault algorithm (only valid in France).
* Has a mental incapacity or language barriers precluding adequate understanding or co operation.
* Has received an investigational drug within the last 28 days preceding Screening Visit or longer if considered to possibly influence the outcome of the current trial.
* Has previously participated in any degarelix trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (52):
- Belgium (4):
  - Hospital St Jan Brugge, Bruges
  - Erasme Hospital, University Clinics of Brussels, Brussels
  - University Hospîtal St-Luc, Brussels
  - University Hospitals Leuven, Leuven
- France (20):
  - CHU Hôpital Sud, Amiens
  - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Hôpital Claude Huriez, Lille
  - Hôpital de la Conception, Marseille
  - Clinique Beausoleil, Montpellier
  - CHU Hôtel-Dieu, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Saint Louis, Paris
  - CHU Pitié Salpétrière, Paris
  - CHU Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Le Milétrie, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital de Rangueil, Toulouse
- Germany (10):
  - Gemeinschaftspraxis Dres. Böhle, Rohde, Bad Schwartau
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Gemeinschaftspraxis - Tagesklinik Dres. Rulf, Langhorst, Erkrath
  - Urologische Gemeinschaftspraxis, Kempen
  - Gemeinschaftspraxis Dres. Rudolph, Wörner, Kirchheim
  - Facharzt für Urologie, Rosenheim
  - Eberhard-Kars-Universität Tübingen, Tübingen
  - Facharzt für Urologie, Wertingen
  - Praxisgemeinschaft f. Onkologie & Urologie, Wilhelmshaven
  - Praxis für Urologie, Zwickau
- Italy (6):
  - Azienda Ospedaliera S. Giuseppe Moscati, Avellino
  - Università degli Studi di Firenze, Bagno A Ripoli (FI)
  - Azienda Policlinico Universitario G. Martino, Messina
  - Ospedale S. Raffaele, Milan
  - Università degli Studi di Padova, Padua
  - Policlinico Univ. Agostino Gemelli, Roma
- Netherlands (5):
  - Twenteborg Ziekenhuis, Almelo
  - Universitair Medisch Centrum Groningen, Groningen
  - Atrium MC Kerkrade, Kerkrade
  - Maatschap Urologie-Diaconessenhuis Leiden, Leiden
  - UMC St.Radboud, Nijmegen
- Spain (7):
  - Complexo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Instituto Valenciano de Oncologia, Valencia

REFERENCES:
- [Derived] Abrahamsson PA, Boccon-Gibod L, Morote J, de Jong IJ, Malmberg A, Neijber A, Albers P. Factors Predicting the Off-treatment Duration in Patients with Prostate Cancer Receiving Degarelix as Intermittent Androgen Deprivation Therapy. Eur Urol Focus. 2017 Oct;3(4-5):470-479. doi: 10.1016/j.euf.2015.12.008. Epub 2016 Jan 22. PMID 28753747
- [Derived] Boccon-Gibod L, Albers P, Morote J, van Poppel H, de la Rosette J, Villers A, Malmberg A, Neijber A, Montorsi F. Degarelix as an intermittent androgen deprivation therapy for one or more treatment cycles in patients with prostate cancer. Eur Urol. 2014 Oct;66(4):655-63. doi: 10.1016/j.eururo.2014.05.037. Epub 2014 Jun 18. PMID 24954791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Degarelix 240 mg / 80 mg
Started | 220 (Randomized participants.)
Safety Analysis Set | 216 (Randomized participants who received ≥1 dose of degarelix.)
Full Analysis Set (FAS), Cycle 1 | 213 (Randomized participants who received ≥1 dose and had ≥1 efficacy assessment.)
FAS, Off-treatment Cycle 1 | 191 (Completed 7 months induction period and were enrolled in the off-treatment period of cycle 1.)
Started Cycle 2 | 35
Started Cycle 3 | 2
Completed | 168 (42, 10, and 0 participants withdrew during Cycles 1, 2, and 3 (i.e. 168 completed the trial).)
Not Completed | 52
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Violation | 5
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 1
Not completed — Miscellaneous reasons | 20

BASELINE CHARACTERISTICS:
Population: FAS, Cycle 1.
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 213
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 212
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  France | 43
  Spain | 24
  Belgium | 26
  Netherlands | 25
  Germany | 63
  Italy | 32
Median Baseline Serum Testosterone Levels [Median (Full Range); unit: ng/mL] | 4.09 [0.1 to 10.0]
Median Baseline Serum Prostate-specific Antigen Levels [Median (Full Range); unit: ng/mL] | 7.9 [0.05 to 61.6]
Baseline EORTC QLQ-PR25 Scores during Cycle 1 [Mean (Standard Deviation); unit: units on a scale] — The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Prostate Module (EORTC QLQ-PR25) assesses urinary, bowel, and sexual symptoms and functioning, and the side-effects of treatment. It consists of 25 questions distributed on these domains (number of items per domain, ranges from x [best possible outcome] to y [worst possible outcome]: urinary symptoms (8, 0-100), bother due to use of incontinence aid (1, 0-100), bowel symptoms (4, 0-100), hormonal treatment-related symptoms (6, 0-100), sexual activity (2, 100-0), and sexual functioning (4, 100-0).
  units on a scale
    Urinary Symptoms | 23.1 (16.0)
    Bother due to Incontinence aid | 18.5 (28.0)
    Bowel Symptoms | 4.05 (9.65)
    Hormonal Treatment-related Symptoms | 7.09 (10.4)
    Sexual Activity | 58.0 (26.8)
    Sexual Functioning | 25.8 (26.7)
Baseline IIEF Scores during Cycle 1 [Mean (Standard Deviation); unit: units on a scale] — The International Index of Erectile Function (IIEF) addresses the relevant domains of male sexual function (i.e. erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction). It consists of the following domains (number of items per domain; ranges from x [worst possible outcome] to y [best possible outcome]: erectile function (6; 1-30), orgasmic function (2; 0-10), sexual desire (2; 2-10), intercourse satisfaction (3; 0-15) and overall satisfaction (2; 2-10).
  units on a scale
    Erectile Function | 7.02 (8.96)
    Orgasmic Function | 2.31 (3.43)
    Sexual Desire | 4.22 (2.26)
    Intercourse Satisfaction | 2.65 (4.2)
    Overall Satisfaction | 5.17 (2.91)

OUTCOME MEASURES:

1. Primary Outcome: Median and Between Participant Variability of Time to Prostate-specific Antigen (PSA) >4 ng/mL During the First Cycle of Intermittent Androgen Deprivation (IAD) After 7 Monthly Injections of Degarelix Induction Treatment
Description: Blood samples for analyses of serum PSA levels were collected at the Screening Visit, and every two months during the course of the trial, and at the End-of-Trial Visit. Analyses were performed using chemiluminometric immunoassay.
Time Frame: Up to 24 months after end of induction period
Population: FAS, Off-treatment Cycle 1, i.e. a subset of all FAS participants who completed the 7 months' induction treatment period of the first cycle and were enrolled in the off-treatment period (of the first cycle) and had at least one efficacy assessment (i.e. PSA or testosterone determination) during the off-treatment period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 191
days | 392 [336 to 448]

2. Secondary Outcome: Percentage Change in PSA Serum Levels From Baseline to the Last Visit of the Induction Period During the First Cycle of IAD
Time Frame: 7 months
Population: FAS, Cycle 1.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 213
percentage of baseline | -90.8 (16.6)

3. Secondary Outcome: Median and Between Participant Variability of Time to Return to Testosterone >0.5 ng/mL (Above Castration Level) During the First Cycle of IAD After 7 Monthly Injections of Degarelix Induction Treatment
Description: Blood samples for analyses of serum testosterone levels were collected at the Screening Visit, Month 4 and 7 of the induction period of Cycle 1 and the corresponding visits of any additional treatment cycles, every two months during the off-treatment period(s), and at the End-of-Trial Visit. Analyses were performed using Liquid-Liquid Extraction and Liquid Chromatography-Mass Spectrometry/Mass Spectrometry.
Time Frame: Up to 24 months after end of induction period
Population: FAS, Off-treatment Cycle 1.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 191
days | 112 [112 to 168]

4. Secondary Outcome: Number of Participants With Testosterone ≤0.5 ng/mL at the Last Visit of the Induction Period During the First Cycle of IAD
Time Frame: 7 months
Population: FAS, Cycle 1.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 213
participants | 210

5. Secondary Outcome: Quality of Life, as Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Prostate Module (EORTC QLQ-PR25), During the Induction Treatment and Off-treatment Periods During the First Cycle of IAD
Description: The EORTC QLQ-PR25 employs a modular approach towards assessing cancer patients´ health-related Quality of Life (QoL) and assesses urinary, bowel, and sexual symptoms and functioning, and the side-effects of hormonal treatment. It consists of 25 questions distributed on six domains (number of items per domain, ranges from x to y: urinary symptoms (8, 0-100), bother due to use of incontinence aid (1, 0-100), bowel symptoms (4, 0-100), hormonal treatment-related symptoms (6, 0-100), sexual activity (2, 0-100), and sexual functioning (4, 0-100). All raw domain scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).
Time Frame: Up to 31 months
Population: FAS, Cycle 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 213
units on a scale
  Urinary Symptoms, End of Induction | 24.5 (18.0)
  Urinary Symptoms, End of Cycle 1 | 21.2 (16.7)
  Bother, End of Induction | 17.9 (29.1)
  Bother, End of Cycle 1 | 31 (34.4)
  Bowel Symptoms, End of Induction | 4.84 (10.2)
  Bowel Symptoms, End of Cycle 1 | 4.98 (8.34)
  Treatment-related Symptoms, End of Induction | 17.6 (14.5)
  Treatment-related Symptoms, End of Cycle 1 | 13.2 (13.0)
  Sexual Activity, End of Induction | 55.1 (27.2)
  Sexual Activity, End of Cycle 1 | 56.7 (26.6)
  Sexual Functioning, End of Induction | 10.9 (17.7)
  Sexual Functioning, End of Cycle 1 | 17.7 (22.6)

6. Secondary Outcome: Sexual Function, as Assessed by the International Index of Erectile Function (IIEF) Scale, During the Induction Treatment and Off-treatment Periods During the First Cycle of IAD
Description: The IIEF scale addresses the relevant domains of male sexual function (i.e. erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction). The IIEF scale is psychometrically sound, and has been linguistically validated in multiple languages. The IIEF scale demonstrates the sensitivity and specificity for detecting treatment-related changes in patients with erectile dysfunction. It consists of the following domains (number of items per domain; ranges from x to y: erectile function (6; 1-30), orgasmic function (2; 0-10), sexual desire (2; 2-10), intercourse satisfaction (3; 0-15) and overall satisfaction (2; 2-10). For all domains, a higher score represents a better sexual function.
Time Frame: Up to 31 months
Population: FAS, Cycle 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 213
units on a scale
  Erectile Function, End of Induction | 3.1 (5)
  Erectile Function, End of Cycle 1 | 5.35 (8.21)
  Orgasmic Function, End of Induction | 0.665 (1.81)
  Orgasmic Function, End of Cycle 1 | 1.76 (3.03)
  Sexual Desire, End of Induction | 2.84 (1.47)
  Sexual Desire, End of Cycle 1 | 3.77 (2.17)
  Intercourse Satisfaction, End of Induction | 0.801 (2.21)
  Intercourse Satisfaction, End of Cycle 1 | 2.01 (3.69)
  Overall Satisfaction, End of Induction | 4.5 (2.9)
  Overall Satisfaction, End of Cycle 1 | 4.97 (3.12)

7. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight During One or More Cycles of Degarelix IAD Treatment
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value during the trial.
Time Frame: Up to 3 x 31 months
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 216
participants
  Systolic blood pressure ≤90 and decrease ≥20 | 4
  Systolic blood pressure ≥180 and increase ≥20 | 13
  Diastolic blood pressure ≤50 and decrease ≥15 | 2
  Diastolic blood pressure ≥105 and increase ≥15 | 8
  Heart rate ≤50 and decrease ≥15 | 4
  Heart rate ≥120 and increase ≥15 | 0
  Body weight decrease of ≥7 percent | 14
  Body weight increase of ≥7 percent | 23

8. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables During One or More Cycles of Degarelix IAD Treatment
Description: This outcome measure included incidence of markedly abnormal changes in safety laboratory values. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value during the trial. ULN=Upper limit of normal.
Time Frame: Up to 3 x 31 months
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg / 80 mg
Number analyzed (Participants) | 216
participants
  S-Alanine Aminotransferase, >3xULN | 2
  S-Alkaline Phosphatase, >3xULN and 25% increase | 1
  S-Aspartate Aminotransferase, >3xULN | 2
  S-Calcium, ≤1.8 mmol/L | 1
  S-Creatinine, ≥177 (µmol/L) | 1
  S-Glutamyltransferase, >3xULN | 1
  S-Potassium, ≥5.8 mmol/L) | 3
  S-Total Bilirubin, >1.5xULN | 1
  S-Urea Nitrogen, >10.7 mmol/L | 24
  S-Sodium, ≤130 mmol/L | 1

ADVERSE EVENTS:
Time Frame: 3 x 31 months.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Groups:
- Degarelix 240 mg / 80 mg: Degarelix 240 mg / 80 mg: For each treatment cycle, a starting dose of 240 mg of degarelix at a concentration of 40 mg/mL was administered on Day 0 as two 120 mg subcutaneous (s.c.) injections in the abdominal region. Thereafter, 6 doses of 80 mg degarelix at a concentration of 20 mg/mL were administered 28 days apart via single s.c. injections.
Arm/Group | Degarelix 240 mg / 80 mg
Serious Adverse Events (participants affected / at risk) | 51/216
Other Adverse Events (participants affected / at risk) | 185/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240 mg / 80 mg (N=216)
Cardiac Failure (Cardiac disorders) | 2
Coronary Artery Stenosis (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 2
Aortic Valve Stenosis (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Diastolic Dysfunction (Cardiac disorders) | 1
Sick Sinus Syndrome (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blindness Transient (Eye disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 2
Inguinal Hernia (Gastrointestinal disorders) | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Tongue Disorder (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Injection Site Oedema (General disorders) | 1
Injection Site Pain (General disorders) | 1
Injection Site Swelling (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Dislocation of Joint Prosthesis (Injury, poisoning and procedural complications) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid Artery Stenosis (Nervous system disorders) | 2
Cerebral Infarction (Nervous system disorders) | 1
Brain Stem Ischaemia (Nervous system disorders) | 1
Cerebral Ischaemia (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Embolic Cerebral Infarction (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Bladder Neck Sclerosis (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal Artery Stenosis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urethral Stenosis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Vascular Pseudoaneurysm (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240 mg / 80 mg (N=216)
Diarrhoea (Gastrointestinal disorders) | 16
Injection Site Pain (General disorders) | 73
Injection Site Erythema (General disorders) | 63
Injection Site Swelling (General disorders) | 48
Injection Site Induration (General disorders) | 31
Fatigue (General disorders) | 30
Oedema Peripheral (General disorders) | 13
Asthenia (General disorders) | 12
Injection Site Pruritus (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 24
Weight Increased (Investigations) | 29
Back Pain (Musculoskeletal and connective tissue disorders) | 15
Headache (Nervous system disorders) | 11
Pollakiuria (Renal and urinary disorders) | 12
Hot Flush (Vascular disorders) | 107
Hypertension (Vascular disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.